CLINICAL TRIAL: NCT04324970
Title: A Prospective Study to Assess Whether the "Tookie Vest for Oncology" Reduces Central Line Fall Out Rate in the Paediatric Oncology Population
Brief Title: Does the "TOOKIE Vest" Reduce Line Fall Out Rate in Children?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R04675
Record Dates: First submitted 2020-03-16; First posted 2020-03-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Childhood Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tookie vest (Experimental): Participant issued with Tookie vest
  Interventions: Device: Tookie Vest

INTERVENTIONS:
Device: Tookie Vest — Tookie Vest

SUMMARY:
The objective of the trial is to assess whether the TOOKIE vest is an effective intervention in reducing line fall out. All oncology patients with a tunneled central line will be approached to participate in this study. Following informed consent they will be issued with a TOOKIE vest.

DETAILED DESCRIPTION:
All oncology patients with a tunneled central line will be approached to participate in this study. Following informed consent they will be issued with a TOOKIE vest. Lines will be studied for the duration they are in situ. This will vary depending on the underlying diagnosis and treatment regime. One hundred central line insertions for oncology patients will be prospectively identified and be given the "TOOKIE Vest" to wear. Data will be collated for each group regarding age, gender, diagnosis, type of central access inserted, duration of line, reason for removal, in cases of infection the infected organism will be documented, date of each fall out.

ELIGIBILITY:
Inclusion Criteria:

* Any child receiving treatment for malignancy at Royal Manchester Children's Hospital
* Patients with a tunnelled central line inserted for treatment of their malignancy

Exclusion Criteria:

• Any child having a portacath inserted as their mode of central access

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-09-06 (Actual); Study Completion 2020-09-06 (Actual)

PRIMARY OUTCOMES:
Central line fall out rate | approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ross Craigie, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No